CLINICAL TRIAL: NCT01790451
Title: The Safety and Efficacy of Irreversible Electroporation for the Ablation of Prostate Cancer Assessed by Procedural Related Side Effects and Post Prostatectomy Histology: A Prospective Human In-Vivo Study.
Brief Title: Safety and Efficacy of Irreversible Electroporation in Ablation of Prostate Cancer in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clinical Research Office of the Endourological Society (Other)
Collaborators: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-252
Record Dates: First submitted 2013-02-08; First posted 2013-02-13 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2014-08

CONDITIONS: Prostate Cancer
Keywords: focal therapy; irreversible electroporation; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- peripheral ablation (Active Comparator): an ablation of the peripheral area of the prostate
  Interventions: Procedure: Irreversible Electroporation
- More central ablation (Active Comparator): an ablation, more centrally, in proximity of the urethra
  Interventions: Procedure: Irreversible Electroporation

INTERVENTIONS:
Procedure: Irreversible Electroporation
  Other Names: Nanoknife

SUMMARY:
Up to 16 patients with confirmed low- or intermediate risk prostate cancer scheduled for a radical prostatectomy will be asked to have the Irreversible Electroporation (IRE) procedure approximately 30 days prior to the prostatectomy. Ablation with IRE will be performed using similar planning criteria, procedure protocol, instruments and software used for brachytherapy, a conventional targeted radiation therapy where radioactive seeds are implanted into prostate tumours. Patients will have an ultrasound of the prostate and the imaging data will be entered into the Planning Software system. The volume of the prostate is measured and a specified ablation zone will be determined. The IRE will be performed under general anaesthetic and the specified zone identified in the planning stage will be ablated. Four IRE electrode needles will be placed into the prostate under ultrasound image guidance. When the needles are in place, electric pulses of one to two minutes duration are used to ablate the specified zone. The total procedure time will be approximately 1 hour. Safety data will be collected and patients will be followed up at 1 week, 2 weeks post IRE, pre- prostatectomy, post prostatectomy and 1 week post prostatectomy. The safety data collection is at 2 weeks post IRE. Before the IRE procedure, patients will have a Magnetic Resonance Imaging (MRI) and Contrast Enhanced Ultrasound (CEUS) of the prostate. The patients will have their scheduled prostatectomy at approximately 30 days after the IRE procedure. Pre-prostatectomy, the ablation zone will be radiologically assessed by a control MRI/CEUS. Post prostatectomy, efficacy of ablation will be determined by histological examination of the prostate by the Pathology Department and measured as complete or incomplete ablation.

The primary outcome is safety as measured by the composite of procedural device and post procedural adverse events, measured with the Common Terminology Criteria for Adverse Events v 4 (CTCAE), Expanded Prostate Cancer Index Composite (EPIC) score, International Prostate Symptom Score (IPSS) or required catheterization time and International Index of Erectile Function (IIEF) and efficacy of ablation determined by histological examination post prostatectomy. Secondary outcomes will be patients procedure satisfaction measured by patient satisfaction questionnaire, post procedural pain management and Visual Analogue Scale (VAS) pain score, time to ambulation, length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with prostate cancer who are indicated to undergo a radical prostatectomy
2. Life expectancy of > 10 years
3. Able to visualize prostate gland adequately on transrectal US imaging during enrolment evaluation
4. No prostate calcification greater than 5 mm
5. Ability of subject to stop anticoagulant and anti-platelet therapy for 7 days prior and 7 days post procedure

Exclusion Criteria:

1. Other Conditions/Status

   1. Bleeding disorder as determined by prothrombin time (PT) > 14.5 seconds, partial thromboplastin time (PTT) > 34 seconds, and Platelet Count < 140/microliter (uL)
   2. Active urinary tract infection (UTI)
   3. History of bladder neck contracture
   4. Anaesthesia Surgical Assignment, category IV or greater
   5. History of inflammatory bowel disease
   6. Concurrent major debilitating illness
   7. Prior or concurrent malignancy
   8. Cardiac History
   9. Implantable cardioverter-defibrillator (ICD) / Pacemaker
2. Prior or current therapies

   1. Biologic therapy for prostate cancer
   2. Chemotherapy for prostate cancer
   3. Hormonal therapy for prostate cancer within 3 months of procedure
   4. Radiotherapy for prostate cancer
   5. Transurethral prostatectomy (TURP), urethral stent
   6. Prior major rectal surgery (except haemorrhoids)
   7. Inability or unwillingness to tolerate temporary cessation of concurrent anticoagulation therapy or anti-platelet drugs for a period of 7days prior to procedure and up to 7 days after procedure

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Safety IRE ablation procedure | 1 year
  To determine if the IRE ablation procedure is safe as measured by the composite number of procedural, device and post procedural adverse events measured with the CTCAE proforma.
Efficacy | 1 year
  To determine if complete ablation of the specified targeted ablation zone is achieved as measured by histopathology assessment.

SECONDARY OUTCOMES:
Side effects | 1 year
  To determine if procedural side effects associated with current treatments for prostate cancer, mainly incontinence, erectile dysfunction and bowel damage are avoided as measured by the validated prostate cancer scores -EPIC, IIEF-5 and IPSS or time of CAD required.
  b) To determine patient satisfaction and comfort measured by Patient Satisfaction Questionnaire, post procedural pain management and pain score, time to ambulation, length of hospital stay.
  c) To determine accurateness of ablation zone detection by MRI/CEUS.
Quality of Life | 1 year
  To determine patient satisfaction and comfort measured by Patient Satisfaction Questionnaire, post procedural pain management and pain score, time to ambulation, length of hospital stay.
Ablation Zone Detection | 1 year
  To determine accurateness of ablation zone detection by MRI/CEUS

CONTACTS AND LOCATIONS:
Locations (1):
- AMC University Hospital, Amsterdam, Netherlands

REFERENCES:
- [Derived] van den Bos W, de Bruin DM, Jurhill RR, Savci-Heijink CD, Muller BG, Varkarakis IM, Skolarikos A, Zondervan PJ, Laguna-Pes MP, Wijkstra H, de Reijke TM, de la Rosette JJ. The correlation between the electrode configuration and histopathology of irreversible electroporation ablations in prostate cancer patients. World J Urol. 2016 May;34(5):657-64. doi: 10.1007/s00345-015-1661-x. Epub 2015 Aug 22. PMID 26296371
- [Derived] van den Bos W, de Bruin DM, Muller BG, Varkarakis IM, Karagiannis AA, Zondervan PJ, Laguna Pes MP, Veelo DP, Savci Heijink CD, Engelbrecht MRW, Wijkstra H, de Reijke TM, de la Rosette JJMCH. The safety and efficacy of irreversible electroporation for the ablation of prostate cancer: a multicentre prospective human in vivo pilot study protocol. BMJ Open. 2014 Oct 29;4(10):e006382. doi: 10.1136/bmjopen-2014-006382. PMID 25354827
- See also: Related Info — http://www.croesoffice.org